CLINICAL TRIAL: NCT00351637
Title: Sublingual Methadone for the Management of Cancer-related Procedure Pain in Inpatients: a Phase II Multicenter, Open Label, Feasibility Study
Brief Title: Sublingual Methadone for the Management of Cancer-related Procedure Pain in Inpatients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study suspended due to low accrual
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20145; 22206
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2012-01-19 (Estimated); Status verified 2012-01

CONDITIONS: Cancer; Pain
Keywords: Sublingual methadone; iatrogenic; treatment related incident breakthrough pain; feasibility study; Phase II/open-label; inpatients; Safety/efficacy; Cancer related breakthrough pain; previously receiving opioids; speak English
MeSH Terms: conditions — Neoplasms; Pain

INTERVENTIONS:
Drug: Sublingual Methadone

SUMMARY:
The purpose of this Phase II study is to determine the feasibility of the dose titration and assessment protocol in the impatient population, in the clinical setting of preventing or managing breakthrough pain, before conducting an appropriately powered phase III study. Thus the primary purpose of this study is to determine the proportion of patients who are successfully titrated to an effective dose of sublingual methadone.

ELIGIBILITY:
Inclusion Criteria:

* Pain due to cancer or its treatment; Controlled baseline pain; episodes of predictable, treatment related pain every day that are 4"/10" in severity or greater, last 10 minutes or longer, or episodes of breakthrough pain not related to cancer treatment, and are responsive to short acting oral opioids such as morphine or hydromorphone; are able to hold a volume of 1.0cc of water under tongue for a 2-minute period; are able to provide written informed consent; are able to fill out the study forms, and are inpatients

Exclusion Criteria:

* Severe underlying respiratory disease such that the investigator is wary about the risk of respiratory failure from modest doses od opioid; prior sensitivity to methadone; currently are being administered methadone; are clinically unstable or have a life expectancy of less than one month making completion of the trial unlikely; and if they do not understand English sufficiently to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
to demonstrate the feasibility of a novel model to assess sublingual methadone to relieve iatrogenic,
treatment related incident breakthrough pain.

SECONDARY OUTCOMES:
to develop a research tool
the Breakthrough Pain Assessment Tool (BPAT)
and to demonstrated proof of concept

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hagen, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Tom Baker Cancer Center, Calgary, Alberta, Canada